CLINICAL TRIAL: NCT07262723
Title: Efficacy and Safety of Levosimendan in Patients With Acute Decompensated Heart Failure: A Real-World Evidence
Brief Title: Levosimendan in Acute Decompensated Heart Failure
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Collaborators: Beacon Pharmaceuticals PLC (Unknown); Pi Research and Development Center, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Anisul Awal, Associate Professor, Department of Cardiology, Chittagong Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59.127.1557.013.19.PG.2025.364
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Decompensated Heart Failure (ADHF)
Keywords: Acute decompensated heart failure (ADHF); Levosimendan; Real-world evidence; Efficacy; Safety; NT-proBNP / pro-BNP levels; Randomized controlled trial (RCT); Electrocardiogram (ECG); Good Clinical Practice (GCP); Declaration of Helsinki; Adverse events
MeSH Terms: interventions — Simendan; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment interventional model. Adults with acute decompensated heart failure will be randomized by computer-generated block randomization (block size six) into two groups. The experimental arm will receive standard guideline-directed care plus levosimendan infusion (0.1 μg/kg/min for 24 hours), while the control arm will receive standard care alone following the 2024 ACC guidelines. The trial is open-label, with both investigators and participants aware of treatment assignments. The primary purpose is treatment, evaluating the efficacy and safety of levosimendan in real-world clinical practice. A total of 332 patients (166 per arm) will be enrolled and followed for 90 days, with assessments at baseline, 6h, 24h, 5 days (or discharge), and 90 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will receive standard guideline-directed care for heart failure plus levosimendan infusion. Levosimendan will be administered as a continuous intravenous infusion at 0.1 μg/kg/min for 24 hours, in addition to standard therapy.
  Interventions: Drug: Levosimendan
- Standard Care (Active Comparator): Participants will receive standard guideline-directed care for heart failure according to the 2024 ACC guidelines. This may include diuretics, vasodilators, inotropes, and other evidence-based therapies as clinically indicated.
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Levosimendan — Levosimendan is a calcium-sensitizing inotrope with vasodilatory effects, enhancing heart contractility without raising oxygen demand and promoting vascular relaxation. In this trial, patients will be randomized to receive either standard care alone or standard care plus levosimendan (0.1 μg/kg/min IV infusion for 24 hours).
  Arms: Intervention Arm
Other: Standard care — Participants will receive standard care for acute decompensated heart failure according to the 2024 ACC Guideline for the Management of Heart Failure. This may include intravenous diuretics, vasodilators, inotropes, renin-angiotensin system inhibitors, beta-blockers, mineralocorticoid receptor antagonists, and SGLT2 inhibitors as clinically indicated.
  Arms: Standard Care

SUMMARY:
Acute decompensated heart failure (ADHF) is one of the major causes of hospitalization and mortality worldwide. Despite advances in medical treatments, managing ADHF remains complex, especially in high-risk populations. Levosimendan, a calcium sensitizer that improves myocardial contractility and reduces complications associated with acute decompensated heart failure, has shown potential in improving outcomes in these patients. The present study aims to evaluate the efficacy and safety of levosimendan in patients with ADHF in a real-world clinical setting.

This pragmatic, multicenter, randomized, controlled trial will include adult patients diagnosed with ADHF in two groups: one receiving levosimendan infusion, and the other receiving standard care for heart failure management, according to the most up-to-date clinical protocols. The study is designed to assess both the efficacy and safety of levosimendan, comparing it with the current standard of care.

The primary endpoint of the study will be a clinical composite outcome measured from the NYHA functional classification of heart failure and patient global assessment. Secondary endpoints will include change in serum pro-BNP levels, clinical outcome of heart failure, changes in dyspnea status, all-cause and cardiac mortality. Safety endpoints, including adverse events, will also be systematically recorded and analyzed. Adverse events will be closely monitored, categorized as either mild, moderate, or severe, and their potential association with the treatment will be assessed.

Data collection will occur at baseline and during subsequent follow-up visits at 6 hours, 24 hours, 5 days (or day of discharge), and 90 days post-treatment. Key efficacy measures will be obtained through clinical evaluations and laboratory tests, including blood pressure, electrocardiogram (ECG) findings, and NT-proBNP serum levels. The statistical analysis will follow an intention-to-treat (ITT) and Per protocol (PP) approach to account for all enrolled patients, ensuring robust and generalizable findings. This study will be conducted in accordance with Good Clinical Practice (GCP) guidelines and ethical standards outlined in the Declaration of Helsinki, prioritizing participant safety and scientific rigor throughout the study.

12 The results of this trial will provide critical insights into the potential benefits of levosimendan for treating ADHF, and could potentially inform clinical decision-making, offering a more effective therapeutic option in managing this life-threatening condition.

DETAILED DESCRIPTION:
INTRODUCTION:

Heart failure (HF) is a clinical syndrome characterized by the reduced capacity of the left ventricle of the heart to pump or fill with blood, often leading to inadequate cardiac output and compensatory mechanisms such as neurohormonal activation and increased left ventricular filling pressures. Globally, HF affects an estimated 64.3 million people, marking it one of the major public health concern. Acute decompensated heart failure (ADHF), a clinical stage of HF, characterized by a rapid deterioration of symptoms and necessitates immediate medical attention. ADHF is particularly associated with high morbidity and mortality rates, significant healthcare utilization, and adverse long-term outcomes. ADHF contributes significantly to hospital admissions, especially among patients with heart failure with reduced ejection fraction (HFrEF). In high-income countries such as the United States and Europe, ADHF accounts for over one million hospitalizations annually. Alarmingly, approximately 24% of these patients are readmitted within 30 days, and 50% experience rehospitalization within six months. The recurrence of HF exacerbations often leads to a worsening prognosis, progressive multiorgan dysfunction, and increased mortality, with one in six patients succumbing within 30 days of hospitalization.

The burden of HF is even more in low- and middle-income countries (LMICs), including Bangladesh, though data is limited. In LMICs, delayed diagnosis, resource limitations, and late-stage presentation exacerbate the challenges of HF management. Bangladesh is experiencing a rising prevalence of cardiovascular diseases, with HF emerging as a leading cause of hospitalization and mortality along with increased life expectancy and aging of the population. Factors such as hypertension, diabetes, coronary artery disease, and rheumatic heart disease contribute significantly to the incidence of HF in the region. The healthcare infrastructure in Bangladesh is often ill-equipped to handle the complex needs of HF patients, with limited access to advanced diagnostic tools, medications, and specialized care. This leads to frequent hospitalizations and poor outcomes for patients with ADHF.

The management of ADHF involves a combination of pharmacological and non-pharmacological strategies aimed at stabilizing the patient, alleviating symptoms, and improving hemodynamic parameters. Diuretics, particularly loop diuretics, are the cornerstone of ADHF treatment, effectively reducing fluid overload. However, diuretics alone do not address the underlying pathophysiology of HF, leaving patients with severe symptoms inadequately managed. Inotropic agents such as dobutamine and dopamine are often employed to enhance cardiac output in more severe cases. Vasodilators like nitroglycerin and nitroprusside are additional options, particularly in patients with hypertension and pulmonary congestion.

Beside these pharmacotherapies, Levosimendan, a calcium-sensitizing inotropic agent, represents a significant advancement in the treatment of ADHF. Unlike traditional inotropes, Levosimendan enhances myocardial contractility without markedly increasing myocardial oxygen consumption, thereby reducing the risk of tachyarrhythmias and ischemic events. Its dual action as an inotrope and vasodilator allows it to improve both cardiac output and systemic vascular resistance, making it particularly effective in patients with severe low-output HF. Clinical evidence suggests that Levosimendan improves symptoms, reduces hospital length of stay, and, in some studies, decreases mortality. Additionally, it's unique mechanism of action and sustained hemodynamic effects-mediated through its active metabolite-offer an extended therapeutic window even after the cessation of infusion.

Despite the promising evidence supporting Levosimendan, its adoption as a standard treatment for ADHF remains limited in Bangladesh. In this context, understanding the efficacy and safety of levosimendan in improving clinical outcomes, reducing rehospitalizations, and mortality in ADHF is important in this country. Hence, the present study will aim to investigate the efficacy and safety of levosimendan in patients with ADHF in Bangladesh.

OBJECTIVES:

Primary objective:

• To investigate the efficacy and Safety of Levosimendan in patients with acutely decompensated heart failure (ADHF).

Secondary objectives:

* To investigate the short-term efficacy of Levosimendan in terms of clinical improvements in patients with ADHF
* To investigate the long-term efficacy of Levosimendan in terms of mortality and hospital readmission in patients with ADHF
* To investigate the adverse events of Levosimendan in patients with ADHF

RATIONALE:

Levosimendan has shown benefits in clinical trials by improving hemodynamics, reducing hospital stay, and enhancing survival in acute heart failure. However, its adoption in guidelines remains inconsistent, particularly in low- and middle-income countries like Bangladesh. Most evidence comes from Western populations, leaving gaps in contextual data for South Asia, where genetic and ethnic variations may affect drug response. Limited real-world evidence exists in Bangladesh, especially compared to other inotropes like dobutamine, and data on long-term outcomes such as mortality and re-hospitalization are scarce. This study aims to generate baseline evidence on the short- and long-term safety and efficacy of Levosimendan in Bangladeshi patients with acute decompensated heart failure.

Drug profile (Levosimendan) Levosimendan is a calcium-sensitizing inotropic agent with vasodilatory properties. Its primary mechanism of action is stabilizing the calcium-troponin C complex in cardiac myocytes, leading to increased myocardial contractility without raising intracellular calcium levels or myocardial oxygen consumption. Additionally, it activates ATP-sensitive potassium (K-ATP) channels in vascular smooth muscle and mitochondria, resulting in systemic and coronary vasodilation. These dual effects improve both myocardial and peripheral perfusion, addressing key hemodynamic abnormalities in ADHF.

The pharmacodynamic profile of levosimendan offers multiple hemodynamic benefits. By enhancing contractility and activating K-ATP channels, it effectively increases cardiac output, reduces pulmonary capillary wedge pressure (PCWP), and lowers systemic vascular resistance (SVR). These actions lead to improved peripheral organ perfusion and symptomatic relief for patients with ADHF. Unlike traditional inotropes such as dobutamine and dopamine, levosimendan does not rely on beta-adrenergic receptor activation or increase intracellular calcium, making it safer for patients with pre-existing arrhythmias or ischemic heart disease. Furthermore, its mitochondrial K-ATP channel activation may provide cytoprotective effects, reducing myocardial injury during ischemic episodes.

Administered intravenously with a typical regimen of a continuous infusion of 0.05-0.2 μg/kg/min for up to 24 hours, levosimendan is immediately bioavailable. It is highly protein-bound (~97-98%), allowing efficient distribution to target tissues. It undergoes hepatic metabolism through conjugation, producing an active metabolite, OR-1896, which has a significantly prolonged half-life of 70-80 hours. This metabolite is primarily excreted via the kidneys and accounts for the drug's sustained hemodynamic effects, which can last for up to 7-9 days after the infusion.

Levosimendan has shown consistent efficacy across several clinical trials. RCTs, such as LIDO, REVIVE, and SURVIVE have highlighted its ability to improve hemodynamic parameters, alleviate symptoms, and reduce hospital length of stay. The drug's safety profile is also notable. Levosimendan is generally well-tolerated, with hypotension, headache, and hypokalemia being the most commonly reported adverse effects. Importantly, it is associated with a lower incidence of tachyarrhythmias compared to traditional inotropes, making it a safer option for patients with ADHF.

Study design The proposed study will be designed as a pragmatic, two-arm, open-labelled, randomized, controlled trial conducted in a real-world clinical setting.

METHODS:

Study setting

* The present study will be conducted in following institutions:
* Chattogram Medical College Hospital, Chattogram, Bangladesh
* National Institute of Cardiovascular Diseases, Dhaka, Bangladesh
* Chattogram Maa-O-Shishu Hospital Medical College Hospital, Chattogram, Bangladesh
* Dhaka Medical College Hospital, Dhaka, Bangladesh
* United Hospital Limited, Dhaka, Bangladesh
* Cox's Bazar Medical College
* Apollo Imperial Hospital & Max Hospital, Chattogram.

Study duration The duration of the present study will be 12 months, from July 2025 to June 2026.

Study population The study population will include adult patients aged over 18 years, who will present with acute decompensated heart failure (ADHF) with a history of left ventricular dysfunction as demonstrated by a left ventricular ejection fraction (LVEF) of less than 40% within the past 12 months (calculated by Simpson's method)

Sample size calculation Final sample is calculated as 166 patients in each arm, a total of 332 patients.

Sampling procedure A purposive sampling technique according to the inclusion and exclusion criteria will be used for recruitment of study participants.

Eligibility criteria Inclusion criteria

* Adult patients (age >18 years)
* Both male and female sex
* Having left ventricular dysfunction, evidenced by a left ventricular ejection fraction <40% within the prior 12 months
* Hospitalized for the treatment of ADHF
* Remained dyspneic at rest despite treatment with intravenous diuretics (NYHA class IV)
* Patients might have received intravenous vasodilators and/or positive inotropic drugs (except amrinone and milrinone), but the infusion rates of these drugs must have remained constant for at least 2 h before entry into the study.

Exclusion criteria

* History of invasive cardiac procedure

  * Cardiac surgery during lifetime within 3 months prior to screening
  * Cardiac revascularization within 3 months prior to screening
  * Left ventricular assist device (LVAD) implantation within 3 months prior to screening
  * A cardioversion within 4 h prior to screening, or
  * Cardiac re-synchronization procedure within 30 days prior to screening)
* Rhythm disorders (e.g. earlier Torsades de Pointes, increased heart rate)
* Severe ventricular outflow obstruction
* Angina within 6 h prior to screening
* Hypotension (a systolic blood pressure <90 mmHg) [Can be included after resuscitation, when SBP will be >90 mmHg by noradrenaline infusion]
* Uncorrected hypokalemia
* CNS disease (e.g. stroke, TIA)
* Respiratory (e.g. COPD exacerbation requiring systematic steroids or intubation)
* Renal insufficiency (e.g. increased serum creatinine clearance rate <15 mL/min)
* Hepatic impairment (e.g. significant increase in liver enzymes, >5x the upper limit of normal)
* Decompensation from active infection eg, sepsis
* Acute bleeding
* Patient required blood transfusion or Severe anemia (hemoglobin <8 g/l)
* Serum potassium concentration <3.5 or >5.4 mmol/l
* Use of amrinone and milrinone prior to screening
* A history of hypersensitivity to levosimendan or any of the excipients
* Intubated or otherwise unable to communicate
* Pregnancy
* Post-partum cardiomyopathy
* Previous participation in a clinical trial with any experimental treatment within the last 30 days

Study procedure

Following steps will be implemented for conducting the present study:

1. Recruitment and training of data collectors
2. Screening and enrollment of the participants
3. Treatment allocation, provision and administration of drugs and
4. Follow up of the participants

Recruitment and training of data collectors For data collection in the present study, one study physician/research assistant will be recruited for each of the study site. After recruitment, the research assistant will be trained on the protocol and data collection procedure of the present study. Two-day training will be arranged and included all the Research assistants and other stakeholders of the study before induction of the data collection.

Participant screening and enrollment Patients admitted to the relevant hospitals will be screened for eligibility in the present study. If the patient meets the inclusion criteria, he/she will be recruited for further study procedure.

Consenting participants The selected individuals will be informed about the aim, procedure and benefit of the study, and written informed consent will be obtained from the patients in their own language [Bengali] by the research assistant working on the trial.

Randomization This study will use block randomization with a block size of six to maintain balanced allocation between the levosimendan and standard care groups. A computer-generated randomization sequence will be prepared and securely stored in opaque envelopes. The sequence will be managed by a third party (Pi Research and Development Center) and provided to the investigator to ensure impartiality and minimize selection bias.

Blinding This study will be conducted as an open labelled trial.

Treatment Allocation Participants will be randomly assigned to one of two groups: the intervention group receiving levosimendan or the control group receiving standard care for heart failure. Treatment will be allocated following eligibility confirmation and baseline assessments.

Intervention Group (standard care+ Levosimendan) Participants in the intervention group, along with standard care for heart failure, will receive levosimendan, administered as a continuous intravenous infusion at a rate of 0.1 μg/kg/min for 24 hours. The drug will be infused through a peripheral vein using a calibrated infusion pump, ensuring precise and controlled administration. The infusion pump will be monitored by trained physicians/nurses to maintain the required dosing rate throughout the treatment period. The participants will be observed for any potential adverse effects during and after the infusion, with continuous monitoring of vital signs to ensure safety.

Control Group (standard care) Participants in the control group will receive standard care for heart failure, which may include intravenous diuretics, vasodilators, inotropes, and other interventions based on the patient's clinical status. The 2024 ACC Guideline for the Management of Heart Failure will be followed for patients' management in the present study. A schematic guideline is provided below according to the guideline is provided below.

1. Initial Assessment Assess severity of congestion and perfusion Identify and address precipitating factors (e.g., ACS, arrhythmias, infections, medications)
2. Decongestion Strategy Administer IV loop diuretics promptly for significant fluid overload

   If diuresis is inadequate:
   * Increase IV loop diuretic dose (frusemide)
   * Add Acetazolamide
3. Continue or Optimize GDMT (It includes 4 groups of drugs) Group 1: Renin-Angiotensin System Inhibition Prefer ARNi (sacubitril/valsartan) for HFrEF

   * If not feasible: Use ACE inhibitor (e.g., enalapril)
   * If ACE inhibitors not tolerated: Use ARB (e.g., valsartan) Group 2: Beta-Blockers Use evidence-based beta-blockers (e.g., carvedilol, bisoprolol) after stabilization Group 3: MRAs Spironolactone or eplerenone if eGFR >30 mL/min and K+ <5.0 mEq/L Group 4: SGLT2 Inhibitors Empagliflozin or dapagliflozin or for all patients
4. Adjunctive Therapies Consider IV vasodilation therapy (nitroglycerin or nitroprusside) for dyspnea relief in absence of hypotension
5. Venous Thromboembolism (VTE) Prophylaxis Administer anticoagulants to prevent VTE (if required)
6. If cardiogenic shock present Use intravenous inotropes (noradrenaline) to maintain systemic perfusion and preserve organ function. Milrinone or amrinone will not be permitted within 24h of randomization.

Dose modification:

The infusion of the study medication (levosimendan) will be stopped if patients experience any of the following conditions to ensure their safety:

If a patient develops symptomatic hypotension, characterized by symptoms such as dizziness, syncope, or signs of inadequate tissue perfusion, the dose of study medication (Levosimendan) will be halved (0.05 μg/kg/min), until the BP is settled (SBP >90 mmHg). If, BP continues to fall or remained unchanged after halving the dose, infusion of Levosimendan will be halted. During this period, noradrenaline can be infused at a dose of 0.2 to 0.4 μg/kg/min, based on best clinical judgement and patient condition to raise the BP. After the SBP rise >90 mmHg, Levosimendan can be re-initiated at the half dose (0.05 μg/kg/min). If, BP remains stable (for 30 minutes), dose of Levosimendan can be increased to 0.1 μg/kg/min. Total infusion of Levosimendan should be completed within 24 (+6) hours.

Additionally, if any serious adverse event (SAE) occurs, which in the investigator's judgment may be related to the study medication, the infusion will be stopped immediately. SAEs can include any significant health event that may require medical intervention and monitoring.

If the infusion is stopped, the patient will be closely monitored, and appropriate medical management will be provided. The decision to modify or discontinue the treatment will prioritize patient safety at all times.

Rescue medication:

In the event that patients develop persistent hypotension or refractory heart failure during the infusion of levosimendan, rescue medication will be administered as necessary. Specifically, intravenous noradrenaline may be used to manage these conditions. The recommended dose of intravenous noradrenaline is 0.2 to 0.4 μg/kg/min, based on best clinical judgement and patient condition.

The decision to administer noradrenaline will be at the discretion of the treating physician, guided by clinical judgment and the patient's response to levosimendan infusion. Patients will be closely monitored for any adverse effects related to the use of rescue medication, and adjustments will be made as needed to ensure optimal patient safety and outcomes.

Follow-up Schedule:

Follow-up Schedule Participants will have follow-up visits at 6 hours, 24 hours, day 5 or discharge, and day 90 (+/- 7 days). Assessments will include vital signs, clinical status, patient-reported outcomes, laboratory and imaging studies, morbidity and mortality data, and adverse event monitoring. Missed visits will be proactively managed via contact and rescheduling.

Discontinuation and Withdrawal Participants may discontinue or withdraw at any time without penalty. Study medication may be discontinued early for safety reasons or per investigator judgment. Discontinuations will be carefully managed to maintain safety and data integrity.

Statistical Analysis:

The primary analysis will be conducted on an intention-to-treat (ITT) population, including all randomized patients who receive at least one dose of the study drug. A per-protocol (PP) analysis will also be performed excluding patients with major protocol deviations. Descriptive statistics will summarize baseline characteristics, using mean and standard deviation for normally distributed continuous variables, median and interquartile range for skewed variables, and frequencies and percentages for categorical variables.

Comparisons of continuous outcomes between treatment groups will be performed using independent Student's t-tests or nonparametric equivalents such as the Mann-Whitney U test, depending on data distribution. Categorical outcomes will be analyzed using Chi-square or Fisher's exact tests. Time-to-event analyses, such as mortality or rehospitalization, will be analyzed using Kaplan-Meier survival curves and compared by log-rank test. Multivariable Cox proportional hazards models may be used to adjust for potential confounders.

Missing data will be handled using appropriate methods, including sensitivity analyses. Statistical significance will be considered at p-values less than 0.05. Statistical analyses will be conducted using standard software such as SPSS or Stata.

Adverse Events Management:

All adverse events (AEs) occurring during the study period will be recorded in detail, including severity, duration, outcome, and relationship to study medication. AEs will be categorized as mild, moderate, or severe. Serious adverse events (SAEs) are defined as those resulting in death, life-threatening conditions, hospitalization or prolongation of hospitalization, significant disability, or congenital anomalies.

Study participants will be closely monitored during and after levosimendan infusion for any signs of adverse reactions. If a patient develops symptomatic hypotension, the levosimendan dose will be reduced by half or discontinued based on clinical judgment. In case of persistent hypotension or refractory heart failure, rescue therapy with intravenous noradrenaline may be initiated.

All SAEs will be immediately reported to the principal investigator and ethical review committee as per regulatory requirements. Appropriate medical intervention and follow-up will be ensured for patients experiencing AEs or SAEs. The study may be paused or stopped if safety concerns arise.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years)
* Both male and female sex
* Having left ventricular dysfunction, evidenced by a left ventricular ejection fraction <40% within the prior 12 months
* Hospitalized for the treatment of ADHF
* Remained dyspneic at rest despite treatment with intravenous diuretics (NYHA class IV)
* Patients might have received intravenous vasodilators and/or positive inotropic drugs (except amrinone and milrinone), but the infusion rates of these drugs must have remained constant for at least 2 h before entry into the study.

Exclusion Criteria:

* History of invasive cardiac procedure

  * Cardiac surgery during lifetime within 3 months prior to screening
  * Cardiac revascularization within 3 months prior to screening
  * Left ventricular assist device (LVAD) implantation within 3 months prior to screening
  * A cardioversion within 4 h prior to screening, or
  * Cardiac re-synchronization procedure within 30 days prior to screening)
* Rhythm disorders (e.g. earlier Torsades de Pointes, increased heart rate)
* Severe ventricular outflow obstruction
* Angina within 6 h prior to screening
* Hypotension (a systolic blood pressure <90 mmHg) [Can be included after resuscitation, when SBP will be >90 mmHg by noradrenaline infusion]
* Uncorrected hypokalemia
* CNS disease (e.g. stroke, TIA)
* Respiratory (e.g. COPD exacerbation requiring systematic steroids or intubation)
* Renal insufficiency (e.g. increased serum creatinine clearance rate <15 mL/min)
* Hepatic impairment (e.g. significant increase in liver enzymes, >5x the upper limit of normal)
* Decompensation from active infection eg, sepsis
* Acute bleeding
* Patient required blood transfusion or Severe anemia (hemoglobin <8 g/l)
* Serum potassium concentration <3.5 or >5.4 mmol/l
* Use of amrinone and milrinone prior to screening
* A history of hypersensitivity to levosimendan or any of the excipients
* Intubated or otherwise unable to communicate
* Pregnancy
* Post partum cardiomyopathy
* Previous participation in a clinical trial with any experimental treatment within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement in Heart Failure Symptoms | From baseline to 5 days after treatment initiation
  Improvement in heart failure symptoms during the first five days of treatment, categorized as improved (moderate or marked improvement at 6 hours, 24 hours, and 5 days without deterioration), unchanged (neither improved nor worsened), or worse (persistent unresponsive symptoms after 24 hours, need for rescue intervention, or moderate/marked worsening).

SECONDARY OUTCOMES:
Safety Outcomes - Adverse Events and Serious Adverse Events | From baseline to 90 days follow-up
  Proportion of patients experiencing treatment-related adverse events and serious adverse events, classified by severity and relationship to study medication, monitored from infusion start until 24 hours post-infusion and at hospital discharge.
Changes in Clinical and Functional Status | From baseline to 90 days follow-up
  Changes in serum pro-BNP, patient global assessment scores, patient perception of dyspnea, Killip classification, and NYHA functional class measured at 24 hours, discharge, 30-day, and 90-day visits.
Hospitalization and Mortality Outcomes | During index hospitalization and up to 90 days post-treatment initiation
  Length of hospital stay; in-hospital mortality; rehospitalizations within 90 days; cardiac mortality and all-cause mortality within 90 days.

CONTACTS AND LOCATIONS:
Locations (6):
- Bangladesh (6):
  - Chittagong Medical College Hospital, Chattogram, Chittagong
  - Chattogram Maa-O-Shishu Hospital Medical College Hospital, Chittagong
  - Apollo Imperial Hospital & Max Hospital, Chittagong
  - Cox's Bazar Medical College, Cox’s Bāzār
  - National Institute of Cardiovascular Diseases, Dhaka
  - United Hospital Limited, Dhaka

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) from this study. This decision is based on institutional policy, local regulatory considerations, and the need to protect participant confidentiality. De-identified data may be considered for sharing in the future upon appropriate request and with approval from the study's ethical review committee, but no prospective data sharing plan is in place at present.